CLINICAL TRIAL: NCT01769079
Title: Withdrawal of Nitrate in Patients With Stable Angina - Multicenter Clinical Trial
Brief Title: Clinical Impact of the Withdrawal of Nitrate in Patients With Stable Angina
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GPPG 08-168
Record Dates: First submitted 2012-10-31; First posted 2013-01-16 (Estimated); Last update posted 2014-01-03 (Estimated); Status verified 2014-01

CONDITIONS: Stable Angina; Myocardial Ischemia; Quality of Life
MeSH Terms: conditions — Angina, Stable; Myocardial Ischemia | interventions — Nitrates; Isosorbide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- oral nitrate (Active Comparator): In nitrate group will be provided the same prescribed dose for this drug. One group remains on nitrate use and other on placebo (same number of pills) use.
  Interventions: Drug: Nitrate
- Placebo (Placebo Comparator): In the placebo group will be given the same dose and frequency prescribed nitrate.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nitrate — Two arms: placebo and nitrate
  Other Names: Isosorbide
  Arms: oral nitrate
Drug: Placebo
  Arms: Placebo

SUMMARY:
Chronic treatment of stable angina with nitrates long and short action is extremely frequent. In clinical practice the most commonly observed is a combination of anti-anginal agents, usually including nitrates fixed in an attempt to improve the quality of life of patients, which is not always met with success.

Numerous questions and problems are seen with chronic use of oral nitrates. From a practical standpoint, some advocate the withdrawal of medication in stable patients, while many physicians still hesitate to withdraw the medication by the lack of definitive information about its consequences. In this sense there is a rationale for the attempted removal of nitrate fixed these patients, although evidence to support this action have not been adequately evaluated.

DETAILED DESCRIPTION:
The Ischemic Heart Disease remains in recent years as a major cause of mortality in most of the world, and also the disease that consumes more resources in health in industrialized countries. The use of fixed nitrate in patients with stable angina is quite common, but there is a scarcity of studies showing the need for this medication in this class pacientes.Este study aims to evaluate the consequences of the withdrawal of fixed nitrate in patients with stable angina class I and II, hemodynamically stable for the past six months, as the frequency and duration of episodes of angina, silent ischemia and functional capacity by exercise testing, 24-hour Holter and measurement of quality of life and adherence to therapy. For this purpose, a randomized blinded multicenter clinical trial was designed to placebo (intervention group) X nitrate (control group) in a follow-up period for 4 months. Both groups will receive three evaluations (baseline, 30 days and 120 days) during follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes, aged 18 years or above, with coronary artery disease documented by angiography or noninvasive test (scintigraphy) with stable angina functional class I or II of the Canadian Cardiothoracic Society (CCS), clinically stable for at least six months, using two or more antianginal agents (betablockers or calcium channel antagonist), among them nitrate fixed.

Exclusion Criteria:

* Patients with residence far from the research center and unable to appropriate follow-up. Patients with decompensated heart failure symptoms or class III or IV New York Heart Association (NYHA), poorly controlled hypertension (BP greater than 160/90 mmHg), patients unable to walk or perform stress test and ECG interpretable. Also excluded were patients in the exercise test pre-randomization present significant alterations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2009-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Time of exercise on treadmill test | 4 months
  Evaluate exercise tolerance, time to onset of ischemia and total duration of exercise by exercise testing in patients with stable angina in withdrawal nitrate fixed.

SECONDARY OUTCOMES:
angina function class and time to ischemia on treadmill test | 4 months
  Evaluate the occurrence of angina and/or worsening of functional class (CCS). Assess exercise tolerance and time to onset of ischemia (clinical and electrocardiographic parameters) and total exercise time, through the exercise test. Rate load silent ischemia through 24-hour Holter. Assess quality of life measured by questionnaire Short-Form 36 and Seattle and adherence to medication. Estimate the impact of the withdrawal of nitrate in the Unified Health System.

CONTACTS AND LOCATIONS:
Overall Officials: Carisi A Polanczyk, MD, ScD, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil